CLINICAL TRIAL: NCT04812587
Title: Effects of Exercise Training on Functional Physical Fitness, Balance and Walking in the Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20180002
Record Dates: First submitted 2021-03-08; First posted 2021-03-23 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-02

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The healthy elderly will be were recruited to participate in this study. All the subjects were independent in basic daily living activities, but at least one or more given assistance in the instrumental IADL assessment (ability to use telephone, shopping, food preparing, housekeeping, laundry, mode of transportation, responsibility for own medications, ability to handle finances). Their age should be ranged between 65 - 81 years.
  Interventions: Behavioral: exercise intervention program
- Comparison group (No Intervention): The healthy elderly will be were recruited to participate in this study. All the subjects were independent in basic daily living activities, but at least one or more given assistance in the instrumental IADL assessment (ability to use telephone, shopping, food preparing, housekeeping, laundry, mode of transportation, responsibility for own medications, ability to handle finances). Their age should be ranged between 65 - 81 years.

INTERVENTIONS:
Behavioral: exercise intervention program — The experimental group will receive a 12-week combined exercise intervention program with extra emphasis on balance, muscle strength, and walking ability which involved two 2-hour sessions once per week.
  Arms: Experimental group

SUMMARY:
This study aimed to determine whether a 12-week combined exercise intervention program with extra emphasis on balance, muscle strength, and walking ability was designed to improve functional fitness, balance, walking speed in community-dwelling older people.

DETAILED DESCRIPTION:
1. Written informed consent must be obtained before any study specific procedures are undertaken.

2. The process of the experiment (brief describe)

1. The 30 participants of the experimental group will be recruited from the "community eldercare service" activities, and this group will receive a 12-week combined exercise intervention program with extra emphasis on balance, muscle strength, and walking ability. The other 30 community-dwelling older people of the comparison group who have been involved in a other regular exercise style will not receive our exercise intervention. The comparison group only receives 2 times measurement at an interval of 12 weeks.
2. Subjects completed medical histories, exercise histories, and information on lifestyles by questionnaire and physical examination before participation in the study to ensure they were free from exclusion criteria. The baseline measurements will be conducted before the exercise intervention.
3. The experimental group will receive a 12-week combined exercise intervention program with extra emphasis on balance, muscle strength, and walking ability which involved two 2-hour sessions per week. The exercise program contained aerobic exercises, activities of balance, coordination exercises, strength training, and walking training.
4. After 12 weeks group exercise, the experimental group will receive the second measurements.

ELIGIBILITY:
Inclusion Criteria:

* Independent in basic daily living activities
* At least one or more given assistance in the instrumental Instrumental Activities of Daily Living (IADL) scale

Exclusion Criteria:

* Diagnosis of neurological disease or heart disease
* Assessment do not suitable resistance exercise training, or cannot perform intense activity by doctor

Ages: 65 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Changes in performance of Physical fitness at 12-week | The assessments will be conducted before, immediately after intervention for the experimental group; two times of these assessments to be at an interval of 12 weeks are conducted for the comparison group
  Senior Fitness test (30-second Chair Stand, 30-second Arm Curl, 2-minute Step, Chair Sit and Reach and 8 Foot Up-and-Go)
Changes in Balance and walking ability at 12-week | The assessments will be conducted before, immediately after intervention for the experimental group; two times of these assessments to be at an interval of 12 weeks are conducted for the comparison group
  One leg standing, Five-repetition sit-to-stand test, Timed up-and-go test and Walking speed test

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiun Liaw, Study Director — Kaohsiung Medical University Department of Physical Therapy Associate Professor
Locations (1):
- Li-Jiun Liaw, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage ,and then share with other researchers after publication